CLINICAL TRIAL: NCT05778461
Title: Efficacy of L-ornithine L-aspartate and Therapeutic Plasma Exchange Versus Plasma Exchange Alone in Lowering Ammonia and Improving Outcomes in Pediatric Acute Liver Failure: A Randomized Controlled Trial
Brief Title: Efficacy of L-ornithine L-aspartate and Therapeutic Plasma Exchange Versus Plasma Exchange Alone in Lowering Ammonia and Improving Outcomes in Pediatric Acute Liver Failure.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-ALF-06
Record Dates: First submitted 2023-02-08; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Liver Failure, Acute
MeSH Terms: conditions — Liver Failure, Acute | interventions — ornithylaspartate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-ornithine L-Aspartate (Experimental): LOLA will be administered via continuous intravenous infusion at a dosage of 0.75g/kg/day for 72h (maximum 30g/day). High volume plasma exchange (2x plasma volume) will be started at least 8 hours after initiation of LOLA, and will be completed within 4-5 hours depending on the volume of exchange. Three consecutive cycles of HVPE will be performed, starting at 8h, 32h and 56h respectively.
  Interventions: Drug: L-ornithine L-Aspartate
- Placebo (Placebo Comparator): Placebo will be administered via continuous infusion for 72h, along with HVPE (2x plasma volume) starting at 8h, 32h and 56h respectively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-ornithine L-Aspartate — LOLA will be administered via continuous intravenous infusion at a dosage of 0.75g/kg/day for 72h (maximum 30g/day). High volume plasma exchange (2x plasma volume) will be started at least 8 hours after initiation of LOLA, and will be completed within 4-5 hours depending on the volume of exchange. Three consecutive cycles of HVPE will be performed, starting at 8h, 32h and 56h respectively.
  Arms: L-ornithine L-Aspartate
Drug: Placebo — Placebo will be administered via continuous infusion for 72h, along with HVPE (2x plasma volume) starting at 8h, 32h and 56h respectively.
  Arms: Placebo

SUMMARY:
Pediatric acute liver failure (PALF) is associated with very high mortality and morbidity with native liver survival varying between 21 to 75%.Hyperammonemia manifesting as hepatic encephalopathy and causing cerebral edema isresponsible for poor neurological outcome in ALF. Ammonia lowering measures have led to improvement in HE and higher native liver survival. L-ornithine L-aspartate (LOLA), a salt of natural amino-acids ornithine and aspartate, is an importantammonia scavenging drug. It acts as a substrate for urea cycle in liver and also converts ammonia to glutamine in perivenous hepatocytes as well as in the muscles.This drug has been shown to reduce ammonia and improve hepatic encephalopathy in cirrhoticadults.However, the issue with this drug is that the glutamine formed can reconvert to ammonia by the action of glutaminase, possibly, the reason why it failed to show decrease in ammonia and improvement in native liver survival in a randomized controlled trial in adult ALF. In western countries, ornithine phenylacetate has been used where ornithine converts ammonia to glutamine and phenylacetate then binds to this glutamine to form phenylacetylgutamine and eliminates it. Therapeutic plasma exchange (TPE), both high volume and standard volume has been shown to improve native liver survival in adults with ALF and is the standard of care in management of ALF and a grade 1 recommendation by all eminent liver societies.TPE leads to decreased ammonia. Although rate of ammonia formation is multiple times higher than rate of ammonia removal by plasmapheresis, this ammonia reduction is an indirect effect of glutamine removal by TPE. Glutamine, thus, acts as a reservoir for clearance of ammonia (in muscles and perivenous hepatocytes).In contrast to adults, the response to therapeutic plasma exchange has not been as encouraging inchildren, yet, most centers continue to use it based on recommendations in adults. Based on the knowledge that LOLA converts ammonia to glutamine and TPE clears glutamine from plasma, the investigators hypothesize that LOLA would act in synergestic way with TPE to lower ammonia levels, resulting in improvement in HE and better native liver survival in pediatric ALF. The goal of this clinical trial is to compare L-ornithine L-aspartate and therapeutic plasma exchange versus plasma exchange alone in lowering ammonia and improving outcomes in patients with pediatric acute liver failure.

DETAILED DESCRIPTION:
Methodology:

- Study population

Pediatric acute liver failure patients aged 5-18 years of age, INR > 2, Hepatic encephalopathy (defined by West Haven criteria) and arterial ammonia >100mcg/dL

Study Design:

Interventional - Placebo controlled RCT.

Allocation: Randomized

Method of randomization: Block randomization using Interactive Web Response System (IWRS) with block size 4

Intervention Model: Parallel Assignment

Masking: Double. Patients and investigators will be blinded to treatment assignments. Both intervention and placebo will be prepared and administered by trial nurse.

- Study period

24 months (Feb 2023-Feb 2025)

-- Sample size

As this is a pilot study, a sample size of 16 patients in each arm will be taken.

* Intervention
* In Intervention Arm 1 LOLA will be administered via continuous intravenous infusion at a dosage of 0.75g/kg/day for 72h (maximum 30g/day). High volume plasma exchange (2x plasma volume) will be started at least 8 hours after initiation of LOLA, and will be completed within 4-5 hours depending on the volume of exchange. Three consecutive cycles of HVPE will be performed, starting at 8h, 32h and 56h respectively. In Control Arm, placebo will be administered via continuous infusion for 72h, along with HVPE (2x plasma volume) starting at 8h, 32h and 56h respectively. Placebo will be procured from the same pharmaceutical company manufacturing LOLA. Patients and investigators will be blinded to treatment assignments. Both intervention and placebo will be prepared and administered by trial nurse.
* STATISTICAL ANALYSIS:
* Primary outcome measure: Mann -Whitney U test
* Secondary outcome measures

  * Fisher's exact test for categorical data
  * Mann-Whitney U test for continuous data
* IBM® SPSS® Statistics 29 will be used for statistical analysis. P<0.05 will be considered as statistically significant.
* Adverse effects
* Stopping rule
* Interim analysis will be done after 16 patients. If significant increase in mortality or worsening grade of encephalopathy is seen in the LOLA arm, trial will be stopped. The trial will also be stopped if any significant safety signals related to the adverse effect profile of the study drug is identified in the interim analysis.

  (c) Expected outcome of the project:

The investigators expect LOLA and therapeutic plasma exchange will act synergistically to lower ammonia more effectively and this lowering of ammonia will lead to better native liver survival among children with acute liver failure.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Acute Liver Failure as defined by PALF-Study Group

  * 5-18 years of age
  * INR > 2
  * Hepatic encephalopathy (defined by West Haven criteria)
  * Ammonia >100mcg/dL

Exclusion Criteria:

* Irreversible neurological injury
* Previous treatment with LOLA within 48 hours before admission.
* Acute kidney injury.
* Acute on chronic liver failure
* Those not giving consent

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in ammonia (baseline to day 3) in the 2 groups | 72 hours

SECONDARY OUTCOMES:
Comparison of proportion of participants dying by Day 7 and Day 14 between two groups | Days 7 and 14
Comparison of proportion of participants requiring liver transplant by Day 7 and Day 14 between two groups | Day 7 and Day 14
Comparison of overall survival at Day 7 and Day 14 between two groups | Days 7 and 14
Comparison of change in grade of encephalopathy assessed by West Haven scale by day 3 and day 7 | Day 3 and Day 7
Comparison of optic nerve sheath diameter measured by ultrasound at 24,48 and 72 hours in the 2 groups | 24 hours, 48 hours and 72 hours
To compare the cumulative requirement of mannitol and propofol in the first 72 hours in the 2 groups | 72 hours
Comparison of plasma and dialysate glutamine levels after first cycle of High Volume Plasma Exchange between two groups | 72 hours
Comparison of number of episodes of clinically raised intracranial pressure in the 2 groups | 72 hours
Compare the adverse events in the 2 groups | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tamoghna Biswas, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: No